CLINICAL TRIAL: NCT01224574
Title: Place Des D-dimères Dans la Prise en Charge Des Patients en Fibrillation Auriculaire : Evaluation de la Valeur prédictive Des D-dimères Sur la Survenue d'événements Thromboemboliques
Brief Title: To Assess the Predictive Value of D-dimer Level on the Occurrence of Cardiovascular Events
Acronym: COAGFAII
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Projet Hospitalier de Recherche Clinique Régional, Direction de la Recherche Clinique
Other Study IDs: AOR 01 029
Record Dates: First submitted 2010-09-13; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fribrillation, cardiovascular events, aging, D-dimer
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No biospecimens are to be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of the study was to assess whether D-Dimer level at entry or an increase of D-Dimer level during the follow-up could predict the occurrence of subsequent cardiovascular events in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Patients will be followed-up every 4 months with clinical assessment and D-dimer blinded measurement.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation

Exclusion Criteria:

* follow-up not possible, poor prognosis within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation encountered in usual care
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2001-01; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mahé, MD,PhD, Principal Investigator — Hopital Lariboisière
Locations (1):
- AP HP, Paris, France

REFERENCES:
- [Background] Mahe I, Drouet L, Simoneau G, Minh-Muzeaux S, Caulin C, Bergmann JF. D-dimer can predict survival in patients with chronic atrial fibrillation. Blood Coagul Fibrinolysis. 2004 Jul;15(5):413-7. doi: 10.1097/01.mbc.0000114440.81125.bd. PMID 15205590
- [Background] Mahe I, Drouet L, Chassany O, Mazoyer E, Simoneau G, Knellwolf AL, Caulin C, Bergmann JF. D-dimer: a characteristic of the coagulation state of each patient with chronic atrial fibrillation. Thromb Res. 2002 Jul 15;107(1-2):1-6. doi: 10.1016/s0049-3848(02)00184-6. PMID 12413581
- [Background] Mahe I, Grenard AS, Joyeux N, Caulin C, Bergmann JF. Management of oral anticoagulant in clinical practice: a retrospective study of 187 patients. J Gerontol A Biol Sci Med Sci. 2004 Dec;59(12):1339-42. doi: 10.1093/gerona/59.12.1339. PMID 15699536
- [Background] Lafuente-Lafuente C, Mahe I, Extramiana F. Management of atrial fibrillation. BMJ. 2009 Dec 23;339:b5216. doi: 10.1136/bmj.b5216. No abstract available. PMID 20032065